CLINICAL TRIAL: NCT03901001
Title: A Randomized Controlled Trial of Adjunctive Sirolimus and Oseltamivir Versus Oseltamivir Alone for Treatment of Influenza
Brief Title: Adjunctive Sirolimus and Oseltamivir Versus Oseltamivir Alone for Treatment of Influenza
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sirolimus influenza/Hui/2019
Record Dates: First submitted 2019-03-30; First posted 2019-04-03 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Influenza
Keywords: respiratory; Mortality; cytokines; chemokines
MeSH Terms: conditions — Influenza, Human | interventions — Sirolimus; Oseltamivir

STUDY DESIGN:
Intervention Model Description: randomized trial into either oseltamivir and adjunctive sirolimus or oseltamivir alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oseltamivir and adjunctive sirolimus (Active Comparator): Sirolimus 1 mg daily and oseltamivir 75 mg bid for 5 days, both given orally. Extension of dosing to 10 days for oseltamivir and the study drug is allowed if there is slow recovery, lack of improvement, or deterioration.
  Interventions: Drug: sirolimus and oseltamivir
- oseltamivir alone (Placebo Comparator): oral oseltamivir 75 mg bid alone for 5 days. Extension of dosing to 10 days for oseltamivir and the study drug is allowed if there is slow recovery, lack of improvement, or deterioration.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: sirolimus and oseltamivir — Sirolimus 1 mg daily and oseltamivir 75 mg bid for 5 days, both given orally. Extension of dosing to 10 days for oseltamivir and the study drug is allowed if there is slow recovery, lack of improvement, or deterioration.
  Arms: oseltamivir and adjunctive sirolimus
Drug: Oseltamivir — oral oseltamivir 75 mg bid alone for 5 days. Extension of dosing to 10 days for oseltamivir and the study drug is allowed if there is slow recovery, lack of improvement, or deterioration.
  Arms: oseltamivir alone

SUMMARY:
Seasonal influenza epidemics are important causes of mortality and morbidity. Cytokine dysregulation, with high levels of pro-inflammatory cytokines, occurs in patients with severe influenza A(H1N1)pdm09 virus infection, A(H5N1) infection, and A(H7N9) infection. We aim to investigate the effects of adjunctive sirolimus in adults hospitalized with influenza A or B infections involving the lower respiratory tract.

DETAILED DESCRIPTION:
The investigators aim to investigate the effects of adjunctive sirolimus in adults hospitalized with influenza A or B infections involving the lower respiratory tract. Patients will be randomized to either oseltamivir and adjunctive sirolimus or oseltamivir alone and assessed with reference to normalization of respiratory status (SaO2 ≥93% or respiratory rate ≤20/min on room air) as the primary endpoint,10 cytokines/chemokines and pro-inflammatory mediator changes, viral clearance, symptom resolution, ICU admission/death, day 28 mortality; safety profiles will also be assessed.

The investigators hypothesize that addition of sirolimus to oseltamivir would improve respiratory status and other endpoints more effectively than oseltamivir alone through reduction of inflammatory responses without affecting viral clearance.

ELIGIBILITY:
Inclusion Criteria:

* influenza A and B virus infections confirmed by PCR and/or immunofluorescence assays, hospitalized for the management of severe manifestations of influenza, initiation of oseltamivir, clinical evidence of lower respiratory tract infection (e.g. shortness of breath, tachypnea, oxygen desaturation, crepitations on auscultation, infiltrations or consolidations on chest radiograph) and written informed consent (by the subjects, or from their next of kin if the subjects are unable to provide written consent at the time of enrollment)

Exclusion Criteria:

* use of other immunosuppressants (e.g. post-chemotherapy, post-transplant, autoimmune diseases) other than systemic corticosteroids
* patients with known immuno-compromised conditions (e.g. active haematological malignancies, HIV/AIDS patients who are on antiretroviral therapy and CD4 cell count < 200)
* pregnancy/lactation
* hepatic failure
* patients with surgery done/planned within 1 month
* patients who have received macrolide antibiotics and NSAID for 1 week prior to enrolment due to their immuno-modulating effects
* patients on drugs that may interact and alter sirolimus level (rifampicin, azole antifungals, phenytoin, diltiazem, verapamil, nicardipine, metoclopramide, phenobarbital, carbamazepine) will be excluded for safety purposes
* Use of investigational anti-influenza antivirals and blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
normalisation of respiratory status | 28 days
  SaO2 ≥93% or respiratory rate ≤20/min on room air

SECONDARY OUTCOMES:
viral ribonucleic acid (RNA) in copies per milliliter | 28 days
  All serially collected samples will be subjected to viral ribonucleic acid (RNA) quantification using quantitative reverse transcription PCR (qRTPCR) targeting the matrix (M)-gene ('viral load')
Interleukin 6 in pg/ml | 10 days
interleukin-8 in pg/ml | 10 days
interleukin 17 in pg/ml | 10 days
Chemokine ligand 9 (CxCL9/MIG) in pg/ml | 10 days
Soluble tumour necrosis factor receptor-1 (sTNFR-1) in pg/ml | 10 days
interleukin 18 in pg/ml | 10 days
CRP in mg/L | 10 days
phospho-p38 and phospho-ERK (activated MAPKs) in mean fluorescence intensity(MFI) | 10 days
phospho-inhibitor kB/IkB (NF-kB) in mean fluorescence intensity(MFI) | 10 days
resolution of symptoms in days | 28 days
  A standard questionnaire will be used to collect baseline and serial clinical data. These include clinical manifestations/complications, symptom severity score, vital signs (e.g. temperature, respiratory rate, oxygen saturation), fever duration, requirements for supplemental oxygen therapy and invasive/non-invasive ventilation, duration of hospitalization, death, and occurrence of adverse events.
ICU admission in days | 28 days
mortality in days | 28 days
Incidence of Treatment-Emergent Adverse Events in numbers | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong